CLINICAL TRIAL: NCT01947491
Title: A Comparison of DFD01 Spray Versus Comp01 Lotion, Vehicle Spray and Vehicle Lotion in Subjects With Moderate Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1205
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DFD01 Spray (Experimental): DFD01 Spray twice daily for 28 days
  Interventions: Drug: DFD01 Spray
- Vehicle Spray (Placebo Comparator): Vehicle Spray twice daily for 28 days
  Interventions: Drug: Vehicle Spray
- Comp01 Lotion (Active Comparator): Comp01 Lotion twice daily for 14 days
  Interventions: Drug: Comp01 Lotion
- Vehicle Lotion (Placebo Comparator): Vehicle Lotion twice daily for 28 days
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: DFD01 Spray
  Other Names: Topical corticosteroid spray
  Arms: DFD01 Spray
Drug: Comp01 Lotion
  Other Names: Topical corticosteroid lotion
  Arms: Comp01 Lotion
Drug: Vehicle Lotion
  Arms: Vehicle Lotion
Drug: Vehicle Spray
  Arms: Vehicle Spray

SUMMARY:
The objectives of this study are to compare the safety of DFD01 Spray to Comp01 Lotion for topical treatment of moderate plaque psoriasis and to compare the efficacy of DFD01 Spray to Placebo Spray for topical treatment of moderate plaque psoriasis after 28 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.
* Subjects with psoriasis involving 10 to 20% BSA, not including the face, scalp, groin, axillae and other intertriginous areas.
* Subjects must have an IGA grade of 3 (moderate) at the Baseline Visit

Exclusion Criteria:

* Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
* Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
* Presence of pigmentation, extensive scarring, or pigmented lesions or sunburn which could interfere with the rating of efficacy parameters.
* History of psoriasis unresponsive to topical treatments.
* History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Horizon Research Group, Inc., Mobile, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Encino Research Center, Encino, California
  - Center for Dematology Clinical Research, Inc., Fremont, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Redwood Dermatology Research, Santa Rosa, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - Colorado Medical Research Center Inc., Denver, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - Florida Academic Center Research and Education, Miami, Florida
  - International Dermatology Research Inc., Miami, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - South Bend Clinic, LLP, South Bend, Indiana
  - Compliant Clinical Research Inc., Olathe, Kansas
  - Dermatology Specialists Research, Louisville, Kentucky
  - Lawrence J. Green, MD, LLC, Rockville, Maryland
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Fran Cook-Bolden, MD, New York, New York
  - DermResearch Center of New York Stony Brook Medical Park, Stony Brook, New York
  - Zoe Diane Draelos, MD, PA, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Haber Dermatology & Cosmetic Surgery, Inc., South Euclid, Ohio
  - Carolina Dermatology of Greenville, PA, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Rivergate Dermatology Clinical Research Center, PLLC, Goodlettsville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - The Center for Skin Research, Houston, Texas
  - Stephen Miller, MD, PA, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- [Derived] Sidgiddi S, Pakunlu RI, Allenby K. Efficacy, Safety, and Potency of Betamethasone Dipropionate Spray 0.05%: A Treatment for Adults with Mild-to-moderate Plaque Psoriasis. J Clin Aesthet Dermatol. 2018 Apr;11(4):14-22. Epub 2018 Apr 1. PMID 29657667

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD01 Spray: DFD01 Spray twice daily for 28 days
  DFD01 Spray
- Vehicle Spray: Vehicle Spray twice daily for 28 days
  Vehicle Spray
- Comp01 Lotion: Comp01 Lotion twice daily for 14 days
  Comp01 Lotion
- Vehicle Lotion: Vehicle Lotion twice daily for 28 days
  Vehicle Lotion
Period: Overall Study
Arm/Group | DFD01 Spray | Vehicle Spray | Comp01 Lotion | Vehicle Lotion
Started | 174 | 87 | 90 | 43
Completed | 166 | 81 | 88 | 38
Not Completed | 8 | 6 | 2 | 5
Not completed — Lost to Follow-up | 5 | 3 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Worsening of condition | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD01 Spray | Vehicle Spray | Comp01 Lotion | Vehicle Lotion | Total
Number analyzed (Participants) | 174 | 87 | 90 | 43 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (14.54) | 50.2 (14.12) | 51.0 (12.75) | 51.6 (12.67) | 50.0 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 36 | 34 | 19 | 152
  Male | 111 | 51 | 56 | 24 | 242
Region of Enrollment [Number; unit: participants]
  United States | 174 | 87 | 90 | 43 | 394

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success According to the Investigator Global Assessment (IGA)
Description: IGA of clear or almost clear
Time Frame: Day 15
Population: Efficacy was only done on DFD01 Spray and Vehicle Spray. Protocol specifically noted no efficacy would be done on comparator or its vehicle.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | DFD01 Spray | Vehicle Spray | Comp01 Lotion | Vehicle Lotion
Number analyzed (Participants) | 174 | 87 | 0 | 0
percentage of patients | 19.0 [13.1 to 24.8] | 2.3 [0.0 to 5.4] |  |
Statistical Analysis 1: Comparison: DFD01 Spray vs Vehicle Spray; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Description: One subject in the betamethasone dipropionate 0.05% group had no post-baseline safety evaluations.
Arm/Group | DFD01 Spray | Vehicle Spray | Comp01 Lotion | Vehicle Lotion
Serious Adverse Events (participants affected / at risk) | 0/173 | 1/87 | 2/90 | 0/43
Other Adverse Events (participants affected / at risk) | 23/173 | 15/87 | 19/90 | 20/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray (N=173) | Vehicle Spray (N=87) | Comp01 Lotion (N=90) | Vehicle Lotion (N=43)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray (N=173) | Vehicle Spray (N=87) | Comp01 Lotion (N=90) | Vehicle Lotion (N=43)
Application Site Pain (General disorders) | 13 (13) | 10 (10) | 13 (13) | 10 (10)
Application Site Pruritis (General disorders) | 10 (10) | 9 (9) | 6 (6) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less